CLINICAL TRIAL: NCT04664491
Title: Effect of Standardized Disease Management on Exacerbation of COPD in Primary Health Care in China: a Multicenter, Adjudicator-Blinded, Parallel, Cluster Randomized Clinical Trial
Brief Title: Effects of COPD Standardized Management on COPD Exacerbation
Acronym: COPD STANDARD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Chen Wang, Principal investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-41-K29; 2020-HX-17/214373 (Other Grant/Funding Number: GlaxoSmithKline)
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Standardized Management; Maintenance Therapy; Follow-Up and Monitoring; Lung Function; COPD Symptoms
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: A parallel, cluster randomized trial
Who Masked: Outcomes Assessor
Masking Description: Statisticians and outcome assessors will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standardized management (Experimental): Patients will be managed according to recommendations in GOLD guideline and China's guidelines for COPD care.
  Interventions: Behavioral: Standardized COPD management
- Usual care (Other): Patients will undergo usual care according to current clinical practice in study sites.
  Interventions: Other: Routine COPD management

INTERVENTIONS:
Behavioral: Standardized COPD management — In standardized management group, patients will receive a multifaceted and integrated disease management that follows recommendations in GOLD 2020 and China Guideline on COPD care. It contains the components below.
  1. Maintenance therapy after initial treatment. In this study, patients' initial therapy is the prescribed inhalers at baseline. Maintenance therapy is the medications (LABA, LAMA, or ICS) prescribed for regular or long-term use after initial therapy.
  2. Long-term follow-up and routine monitoring of symptoms measured by CAT, mMRC and SGRQ.
  3. Regular pulmonary function testing for lung function monitoring
  4. Strengthened COPD education
  5. Behavioral modification, eg. encouragement of influenza/pneumococcal vaccination, providing smoking cessation counseling and pulmonary rehabilitation.
  Other Names: COPD management according to GOLD and China's guidelines for COPD care
  Arms: Standardized management
Other: Routine COPD management — Patients will undergo usual care according to current clinical practice in study sites. Usual care is the routine care provided to patients. Prescription and dispense of medicine for COPD initial and maintenance therapy will be at the discretion of doctors.
  Arms: Usual care

SUMMARY:
This is a multi-center, parallel-group,cluster randomised trial involving secondary hospitals across China. The objective is to evaluate the effect of COPD on reducing moderate-to-severe exacerbations during 12 months follow-up in primary-level medical institutions.

DETAILED DESCRIPTION:
COPD is the most common chronic respiratory disease in China. An effective and standardized condition management strategy is urgently needed to prevent acute exacerbation, improve the quality of life, and avoid premature death due to COPD. COPD management is mainly performed in community-level health institutions. Implementing COPD standardized management in primary care will help improve the level of COPD prevention and treatment in China.

The investigators will carry out a multicenter, adjudicator-blinded, parallel, cluster randomized clinical trial. An estimated number of 96 secondary hospitals across the country will be involved. Each hospital plans to enroll 36 patients with COPD. The hospitals will be randomly allocated into standardized management (SM) group and control group. In SM group, standardized COPD management based-on guidelines will be delivered to patients, including inhaler use for initial and maintenance therapy, regular follow-up, long-term monitoring of lung function and respiratory symptoms, patient education, and favorable lifestyle changes. In control group, patients will receive routine care as usual. In both groups, moderate and severe exacerbations will be collected within 12 months follow-up after randomization. Group difference in annual exacerbation rate will be examined to evaluate the effect of standardized management of COPD on acute exacerbation of COPD in primary care.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥40 years
2. Post-bronchodilator FEV1/FVC <70%
3. Baseline CAT score ≥10 or history of exacerbation in previous 12 months, defined as any use of oral antibiotics and/or oral or nebulized corticosteroids for increased cough, sputum and dyspnea, or exacerbation requiring hospitalization/ emergency admission.
4. Local residents who live nearby and can be followed up throughout study period
5. Written informed consent

Exclusion Criteria:

1. Pregnancy, breastfeeding, or potential pregnancy
2. Primary diagnosis of asthma
3. Having severe cognitive dysfunction
4. Severely ill with less than 12-month life expectancy
5. Patients with alcohol abuse history are excluded as alcoholic individuals may have low adherence to the study. Alcohol abuse is defined as an average alcohol intake >80 g per day within recent two weeks, or daily intake of ≥40 g alcohol in men, and ≥20 g alcohol in women for more than 5 years.
6. Have participated in similar trials or are undergoing other clinical trials
7. Refuses or unable to give informed consent
8. Plan to move
9. Contraindicated to maintenance medicine.
10. Unstable cardiovascular conditions (e.g., angina, myocardial infarction, ascending aortic aneurysm) that may prevent patients performing spirometry.
11. Relative contraindications to spirometry, including current pneumothorax or planning to undergo thoracic/abdominal, ophthalmic or brain surgeries within next 6 months.
12. Comorbid lung disease including bronchiectasis and tuberculosis, or undergoing anti-tuberculosis treatment
13. Recent exacerbation treated with antibiotics and/or oral or nebulized corticosteroids within 30 days prior to enrolment.
14. Exacerbation requiring emergency admission or hospitalization within 30 days prior to enrolment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3456 (Estimated)
Dates: Start 2023-02-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | 12 months from baseline
  The primary outcome is annual rate of moderate and severe exacerbation, which will be identified from medical records on the HIS system and patient report at 6 and 12 months assessments

SECONDARY OUTCOMES:
Exacerbation events | 12 months from baseline
  Time to first moderate exacerbation in days, time to first severe exacerbation in days, time to first exacerbation-related hospitalization in days, time to first exacerbation-related emergency admissions in days, time elapsed from patient enrollment until first admission for acute exacerbation in days
Hospital readmissions | 12 months from baseline
  Number of readmissions within 30 days after discharge, time to first readmission within 30 days after discharge in days, number of readmissions within 90 days after discharge, time to first readmission within 90 days after discharge in days
Hospital stay | 12 months from baseline
  Average length of hospital stay in days
Healthcare cost | 12 months from baseline
  Total COPD-related health care cost in rmb
Lung function change | 12 months from baseline
  Change in FEV1 from baseline to 12 months in liter
Symptom change | 12 months from baseline
  Units on SGRQ-C score change from baseline to 12 months, units on CAT score change from baseline to 12 months, units on mMRC score change from baseline to 12 months
Patients' care-seeking behaviors | 12 months from baseline
  Number of patients' contacting physicians for medical advice, number of patients' hospital visits to seek care
Patients' adherence to treatment | 12 months from baseline
  Time of patients' adherence to inhaler medication use in days

OTHER OUTCOMES:
Safety and adverse event | 12 months from baseline
  Number of patients with pneumonia caused by ICS-containing treatment, number of patients with tobacco cessation related adverse events, number of patients with pulmonary rehabilitation related adverse events, number of patients with flu vaccination related adverse events, number of patients with pneumonia vaccination related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Chen Wang, MD, Ph.D, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khakban A, Sin DD, FitzGerald JM, McManus BM, Ng R, Hollander Z, Sadatsafavi M. The Projected Epidemic of Chronic Obstructive Pulmonary Disease Hospitalizations over the Next 15 Years. A Population-based Perspective. Am J Respir Crit Care Med. 2017 Feb 1;195(3):287-291. doi: 10.1164/rccm.201606-1162PP. No abstract available. PMID 27626508
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] Wang C, Xu J, Yang L, Xu Y, Zhang X, Bai C, Kang J, Ran P, Shen H, Wen F, Huang K, Yao W, Sun T, Shan G, Yang T, Lin Y, Wu S, Zhu J, Wang R, Shi Z, Zhao J, Ye X, Song Y, Wang Q, Zhou Y, Ding L, Yang T, Chen Y, Guo Y, Xiao F, Lu Y, Peng X, Zhang B, Xiao D, Chen CS, Wang Z, Zhang H, Bu X, Zhang X, An L, Zhang S, Cao Z, Zhan Q, Yang Y, Cao B, Dai H, Liang L, He J; China Pulmonary Health Study Group. Prevalence and risk factors of chronic obstructive pulmonary disease in China (the China Pulmonary Health [CPH] study): a national cross-sectional study. Lancet. 2018 Apr 28;391(10131):1706-1717. doi: 10.1016/S0140-6736(18)30841-9. Epub 2018 Apr 9. PMID 29650248
- [Derived] Dong F, Su R, Ren Y, Huang K, Li W, Yang L, Li X, Hu X, Ye T, Jin D, Yang T, Jones PW, Wang C. Real-world effectiveness study of guideline-directed COPD STANDARDized management in patients with chronic obstructive pulmonary disease: a cluster randomised trial design. BMJ Open Respir Res. 2025 Jul 7;12(1):e002768. doi: 10.1136/bmjresp-2024-002768. PMID 40623795
- See also: GOLD guidelines — http://www.goldcopd.org